CLINICAL TRIAL: NCT03213652
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice)- Phase 2 Subprotocol of Ensartinib in Patients With Tumors Harboring ALK or ROS1 Genomic Alterations
Brief Title: Ensartinib in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With ALK or ROS1 Genomic Alterations (A Pediatric MATCH Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01243; NCI-2017-01243 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621F (Other: Children's Oncology Group); APEC1621F (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Malignant Solid Neoplasm; Recurrent Ependymoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Hepatoblastoma; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Glioma; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Primary Central Nervous System Neoplasm; Recurrent Rhabdoid Tumor; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Refractory Ependymoma; Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Refractory Hepatoblastoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Germ Cell Tumor; Refractory Malignant Glioma; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Primary Central Nervous System Neoplasm; Refractory Rhabdoid Tumor; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma; Wilms Tumor
MeSH Terms: conditions — Ependymoma; Neuroectodermal Tumors, Primitive, Peripheral; Hepatoblastoma; Histiocytosis, Langerhans-Cell; Glioma; Medulloblastoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Central Nervous System Neoplasms; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Wilms Tumor | interventions — Specimen Handling; Biopsy; ensartinib; Magnetic Resonance Spectroscopy; Nuclear Medicine Department, Hospital; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ensartinib) (Experimental): Patients receive ensartinib PO QD on days 1-28. Cycles repeat every 28 days for 2 years (up to 26 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, CT scan, MRI, PET scan, radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Ensartinib; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Procedure: Radionuclide Imaging; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo a bone marrow aspiration and/or biopsy
Procedure: Bone Scan — Undergo a bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ensartinib — Given PO
  Other Names: X 396; X-396; X396
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Undergo a PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Radionuclide Imaging — Undergo radionuclide imaging
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Procedure: X-Ray Imaging — Undergo an x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II Pediatric MATCH treatment trial studies how well ensartinib works in treating patients with solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with ALK or ROS1 genomic alterations that have come back (recurrent) or does not respond to treatment (refractory) and may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Ensartinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with ensartinib with advanced solid tumors (including central nervous system [CNS] tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor ALK or ROS1 fusions or that harbor ALK missense mutations.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with ensartinib with advanced solid tumors (including CNS tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor ALK or ROS1 fusions or that harbor ALK missense mutations.

II. To obtain information about the tolerability of ensartinib in children with relapsed or refractory cancer.

III. To provide preliminary estimates of the pharmacokinetics of ensartinib in children with relapsed or refractory cancer.

EXPLORATORY OBJECTIVES:

I. To evaluate other biomarkers as predictors of response to ensartinib and specifically, whether tumors that harbor different missense mutations or fusions (including the crizotinib resistant F1174L ALK variant) will demonstrate differential response to ensartinib treatment.

II. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive ensartinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days for 2 years (up to 26 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI), positron emission tomography (PET) scan, radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC//NCI-2017-01251 and must have been given a treatment assignment to Molecular Analysis for Therapy Choice (MATCH) to APEC1621F/NCI-2017-01243 based on the presence of an actionable mutation as defined in APEC1621SC/ NCI-2017-01251
* Patients must be >= than 12 months and =< 21 years of age at the time of study enrollment.
* Patients must have a body surface area >= 0.5 m^2 at enrollment
* Patients must have radiographically measurable disease at the time of study enrollment. Patients with neuroblastoma who do not have measurable disease but have iobenguane (MIBG) positive (+) evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on a standard MRI or CT

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age

  * Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil counts [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial none marrow (BM) radiation

    * Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to ensartinib; prior treatment with other ALK inhibitors is permitted given that at least 5 half-lives or 21 days have elapsed since therapy discontinuation, whichever is greater
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days prior to enrollment)
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) (within 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 (within 7 days prior to enrollment) or a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age 1 to < 2 years: maximum serum creatinine 0.6 mg/dL for male and 0.6 mg/dL for female
  * Age 2 to < 6 years: maximum serum creatinine 0.8 mg/dL for male and 0.8 mg/dL for female
  * Age 6 to < 10 years: maximum serum creatinine 1 mg/dL for male and 1 mg/dL for female
  * Age 10 to < 13 years: maximum serum creatinine 1.2 mg/dL for male and 1.2 mg/dL for female
  * Age 13 to < 16 years: maximum serum creatinine 1.5 mg/dL for male and 1.4 mg/dL for female
  * Age >= 16 years: maximum serum creatinine 1.7 mg/dL for male and 1.4 mg/dL for female
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment) (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL (within 7 days prior to enrollment)
* Patients must be able to swallow intact capsules
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study because there is currently no available information regarding human fetal or teratogenic toxicities; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study treatment and for one week after the last dose of ensartinib
* Concomitant medications

  * Corticosteroids: patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Investigational drugs: patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible
  * Anti-GVHD agents post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
  * CYP3A4 agents: patients who are currently receiving drugs that are strong inducers or strong inhibitors of CYP3A4 are not eligible; strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study

    * Note: CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years from study entry
  A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system (CNS) tumors).

SECONDARY OUTCOMES:
Percentage of patients experiencing grade 3 or higher adverse events | Up to 2 years from study entry
  Percentage of patients experiencing grade 3 or higher adverse events will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All patients who receive at least one dose of protocol therapy will be considered in the evaluation of toxicity.
Progression free survival (PFS) | Up to 6 months from study entry
  The Kaplan-Meier method will be used to estimate the 6 month PFS. PFS is defined as time from initiation of protocol treatment to disease progression, recurrence, death from any cause, or date of last contact.
Pharmacokinetic (PK) parameters | Pre-dose, 1, 2, 4, 6-8, and 20-24 hours post day 1 dose and pre-dose, 1, 2, 4, and 6-8 hours post day 28 dose of cycle 1
  A descriptive analysis of PK parameters will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters. The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).

OTHER OUTCOMES:
Biomarkers as predictors of response to ensartinib | Up to 4 years
  Descriptive analysis will be performed and will be summarized with simple summary statistics.
Changes in tumor genomic profile | Up to 4 years
  Approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid will be explored. Descriptive analysis will be performed and will be summarized with simple summary statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith S Irwin, Principal Investigator — Children's Oncology Group
Locations (126):
- United States (122):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Perth Children's Hospital, Perth, Western Australia, Australia
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Baranowska-Kortylewicz J, Kortylewicz ZP, McIntyre EM, Sharp JG, Coulter DW. Multifarious Functions of Butyrylcholinesterase in Neuroblastoma: Impact of BCHE Deletion on the Neuroblastoma Growth In Vitro and In Vivo. J Pediatr Hematol Oncol. 2022 Aug 1;44(6):293-304. doi: 10.1097/MPH.0000000000002285. Epub 2021 Sep 6. PMID 34486544

DOCUMENTS (1):
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT03213652/ICF_000.pdf